CLINICAL TRIAL: NCT04873011
Title: The Effect of Quinine Hydrochloride on Hedonic Food Intake, Appetite-related Sensations and Gastrointestinal Hormone Release in Overweight Female Subjects
Brief Title: Effect of Quinine Hydrochloride in Overweight Population on Food Intake, Hunger and Gut Peptide Release
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: QOW
Record Dates: First submitted 2021-04-29; First posted 2021-05-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Quinine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quinine hydrochloride (Experimental): The bitter tastant, quinine hydrochloride, will be acutely infused via a nasogastric feeding tube into the stomach. 320 mg of quinine hydrochloride is dissolved in 10 mL of water and all is infused.
  Interventions: Drug: Quinine Hydrochloride
- Placebo (Placebo Comparator): 10 mL of water is infused via a nasogastric feeding tube into the stomach.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quinine Hydrochloride — After a stabilization period of 20 minutes and 10 minutes after the first blood collection, 10 mL of the quinine hydrochloride solution will be infused into the stomach in a randomized, double-blinded fashion
  Arms: Quinine hydrochloride
Drug: Placebo — After a stabilization period of 20 minutes and 10 minutes after the first blood collection, 10 mL of water will be infused into the stomach in a randomized, double-blinded fashion
  Arms: Placebo

SUMMARY:
The worldwide increase in the prevalence of obesity is a cause of great concern. Pharmacological treatment options are being explored at the moment with a major focus on the hormones produced by the gastrointestinal tract which regulate hunger and satiation/satiety. Modulating the release of these hormones via bitter substances reduced appetite-related sensations and gastrointestinal motility in lean female volunteers.

Intragastric administration of a quinine-solution has shown to decrease hunger sensations in healthy female volunteers. Now, we want to examine whether this effect is still seen in an overweight female population.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of acute administration of quinine hydrochloride on the consumed milkshake volume, gastrointestinal hormone levels, appetite-related sensations and whole blood glucose levels in overweight female individuals.

This study is a randomized, placebo-controlled, double blinded, cross-over study. Forty healthy overweight females will be recruited. An acute dose of 320 mg of quinine hydrochloride is administered as a solution via a nasogastric feeding tube. Blood samples will be collected at regular time points to measure gastrointestinal hormone release and whole blood glucose levels. Appetite related sensations will be scored at regular time points on visual analogue scales.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female between 18 and 65 years of age.
* Subject has a BMI between 25 and 30 kg/m² and has a stable body weight for at least 3 consecutive months at the start of the study and keeps a stable weight during the study visits.
* Women of child-bearing age agree to apply during the entire duration of the trial a highly effective method of birth control, which is defined as those which result in a low failure rate (i.e., less than 1% per year) when used constantly and correctly such as implants, injectables, combined oral contraceptive method, or some intrauterine devices (IUDs), sexual abstinence, or vasectomized partner. Women of non-childbearing potential may be included if surgically sterile (tubal ligation or hysterectomy) or postmenopausal with at least 2 year without spontaneous menses.
* Subject understands the study procedures and agrees to participate in the study by giving written informed consent.

Exclusion Criteria:

* Subject is under age of legal consent, male, pregnant or breastfeeding.
* Subject with a BMI ≤ 25 kg/m² or BMI ≥ 30 kg/m².
* Subject has current symptoms or a history of gastrointestinal or other significant somatic or psychiatric diseases or drug allergies.
* Subject is currently following a weight loss diet or other treatment for obesity.
* Subject has diabetes.
* Subject has a significant heart, lung, liver or kidney disease.
* Subject has a QT-interval > 450 ms.
* Subject has any history of a neurological disorder.
* Subject has a history of abdominal surgery. Those having undergone a simple appendectomy more than 1 year prior to the screening visit may participate.
* Subject has retinopathy.
* Subject suffers from psoriasis.
* Subject has porphyria.
* Subject has a hematologic disorder (e.g. hemolysis, thrombocytopenia).
* Subject shows abnormal eating behavior or has a history of an eating disorder.
* History or current use of drugs that can affect glycaemia, gastrointestinal function, motility or sensitivity or gastric acidity.
* History or current use of centrally acting medication, including antidepressants, antipsychotics and/or benzodiazepines (in the last year before screening visit).
* Subject consumes excessive amounts of alcohol, defined as >14 units per week.
* Subject is currently (defined as within approximately 1 year of the screening visit) a regular or irregular user (including "recreational use") of any illicit drugs (including marijuana) or has a history of drug (including alcohol) abuse. Further, patient is unwilling to refrain from the use of drugs during this study.
* High caffeine intake (> 4 cups of coffee daily or equivalent).
* Inability or unwillingness to perform all of the study procedures, or the subject is considered unsuitable in any way by the principal investigator.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female volunteers are lingually more sensitive for the bitter taste compared to males. There are indications that also in the gut, the response is stronger in female volunteers than men.
Enrollment: 40 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2025-10-29 (Estimated); Study Completion 2025-10-29 (Estimated)

PRIMARY OUTCOMES:
To detect changes in consumed milkshake volume after acute administration of quinine hydrochloride compared to placebo. | 60 minutes after quinine hydrochloride or placebo infusion
  Hedonic food intake will be assessed using a chocolate milkshake drinking task. Subjects are instructed to drink ad libitum from a chocolate milkshake until fully satiated. The milkshake will be weighted before and after the experiment. 1 g of chocolate milkshake = 1 kcal.

SECONDARY OUTCOMES:
To detect changes in the release of gastrointestinal hormones after acute administration of quinine hydrochloride compared to placebo. | First sample 10 min prior to administration. Followed by collections every 10 minutes after administration for a period of 90 minutes.
  Gastrointestinal hormone release will be measured in plasma samples collected at regular time points to assess the release of ghrelin, motilin and insulin.
To detect changes in appetite-related sensations after acute administration of quinine hydrochloride compared to placebo. | all appetite-related sensations will be scored every 10 minutes for a period of 110 minutes, starting 20 minutes before quinine or placebo infusion and ending 90 minutes after administration
  Hunger, prospective food consumption, satiety, fullness, bloating, belching, cramps and pain will be scored by the subjects on visual analog scales of 100 mm.
To detect changes in whole blood glucose levels after acute administration of quinine hydrochloride compared to placebo | First sample 10 min prior to administration. Followed by collections every 10 minutes after administration for a period of 90 minutes.
  Whole blood glucose levels will be measured at regular time points with a blood glucose meter.

CONTACTS AND LOCATIONS:
Locations (1):
- TARGID, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No